CLINICAL TRIAL: NCT02916134
Title: Conservative Versus Operative ManageMent of Acute Uncomplicated Appendicitis
Acronym: COMMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Arnold Hill, Professor of Surgery, Beaumont Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/59
Record Dates: First submitted 2016-08-29; First posted 2016-09-27 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Operative Intervention (Active Comparator): Laparoscopic +/- open appendicectomy, with antibiotics at induction and 3 further doses of intravenous antibiotics. Co-amoxiclav, or cefuroxime and metronidazole if previous rash-allergy to penicillin.
  Interventions: Procedure: Laparoscopic +/- Open Appendicectomy
- Antibiotic Treatment (Experimental): Intravenous antibiotics until clinical improvement and then 5 further days of oral antibiotics. Co-amoxiclav, or if rash-allergy to penicillin, cefuroxime and metronidazole.
  Interventions: Drug: Antibiotic treatment

INTERVENTIONS:
Procedure: Laparoscopic +/- Open Appendicectomy — Laparoscopic +/- open appendicectomy , with antibiotics at induction (intravenous co-amoxiclav 1.2g, or if penicillin allergic, cefuroxime 1.5g + metronidazole 500mg ), followed by 3 further intravenous doses of the same antibiotic. If a perforation is identified at the time of surgery, microbiology will be contacted regarding choice and duration of of antibiotic.
  Arms: Operative Intervention
Drug: Antibiotic treatment — Intravenous co-amoxiclav 1.2g three times daily, then 625mg, orally three times daily. If penicillin allergic, intravenous cefuroxime 1.5g three times daily + metronidazole 500mg three times daily, then oral cefuroxime 500mg twice daily + oral metronidazole 400mg three times daily.
  The patient will receive inpatient intravenous antibiotics until sufficient clinical improvement is noted by the surgical team, who will be assessing the patient twice daily. After discharge the patient will receive 5 further days of oral antibiotics.
  Arms: Antibiotic Treatment

SUMMARY:
This study aims to compare antibiotic treatment versus surgery for patients with uncomplicated appendicitis.

DETAILED DESCRIPTION:
The study will include patients aged 16 and over, with a first admission with right iliac fossa pain and a raised white cell count or C-reactive protein. Patients will be randomised electronically in a 1:1 ratio either to undergo emergency appendectomy or to receive intravenous antibiotics as an inpatient, until clinical and biochemical improvement is observed, followed by outpatient oral antibiotics. Those who have surgery will have 3 post-operative doses of intravenous antibiotics, unless perforation was identified at the time of surgery, in which case, microbiology will be contacted to advise regarding antibiotic choice and duration. Follow-up by telephone interview will be at 1 week, 1, 3 and 12-month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Right iliac fossa pain
* 1st episode in the past 1 year
* Raised WCC or CRP
* Fluent in English

Exclusion Criteria:

* History of inflammatory bowel disease or appendectomy
* B-HCG positive
* Significant co-morbidities
* Complicated appendicitis as proven by ultrasound, CT or MRI
* Anaphylaxis to penicillin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2019-12-08 (Actual)

PRIMARY OUTCOMES:
Successful treatment of appendicitis | 1 year post enrollment
  Successful treatment is defined as the resolution of appendicitis resulting in discharge from the hospital and no recurrent appendicitis during the one-year follow-up. The number of patients requiring surgery for appendicitis in the non-operative group will be measured.

SECONDARY OUTCOMES:
Recurrence of appendicitis | 1 year post enrollment
  Confirmed appendicitis occurring after discharge and within one year of enrolment. The number of patients with appendicitis confirmed on either imaging or pathology will be measured.
Clostridium difficile infection | 1 year post enrollment
  Confirmed symptomatic clostridium difficile infection occurring within one year of enrolment. Any patient who presents with diarrhea during the follow-up period or reports diarrhea during assessment with the follow-up questionnaire will be asked to provide a stool sample which will be tested for clostridium difficile toxins.
Need for re-admission or repeat imaging | 1 year post enrollment
  Recurrence or non-resolution of abdominal pain requiring re-admission or re-imaging after discharge and within one year of enrolment. The number of patients who need to be re-admitted to hospital for abdominal pain or require ultrasound, MRI or CT for investigation of abdominal pain during the one year follow-up will be measured.
Quality of life Questionnaire taken over the year after recruitment | 1 year post enrollment
  Quality of life will be measured in both treatment groups at 1 week, 1 month, 3 months and 1 year post enrolment. Quality of life will be measured using the EQ-5D-3L validated quality of life questionnaire.
Complication of treatment | 1 year post enrollment
  Complications of treatment including surgical site infection, abscess formation and ongoing pain will be measured.
Cost evaluation | 1 year post enrollment
  Associated cost will be evaluated in the antibiotics only, surgery and recurrence groups

CONTACTS AND LOCATIONS:
Overall Officials: Arnold K Hill, Principal Investigator — Beaumont Hospital
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No